CLINICAL TRIAL: NCT02834988
Title: The Validity of Sentinel Lymph Node Dissection (SLND) in Patients With Apparent Early Stage Endometrial Cancer (EC)
Brief Title: Sentinel Lymph Node Dissection (SLND) in Patients With Apparent Early Stage Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Other Study IDs: 20151012
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; Sentinel Lymph Node Dissection; SLND
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- SLND Patients: Patients scheduled to have their sentinel lymph nodes removed, as part of standard of care.

SUMMARY:
The investigators hypothesize that SLND (unlike lymphadenectomy) decreases complications such as hemorrhage, lower extremity lymphedema and lymphocyst formation while enhancing quality of life in EC patients with low risk for nodal involvement.

The investigators also hypothesize that SLND is an effective method of staging these patients. Studies have shown that SLN mapping identifies positive lymph nodes in women with newly diagnosed EC and this prognostic information obtained from SLND could guide selection of adjuvant treatment and improve overall survival.

Using SLND as an alternative to lymphadenectomy may also have additional medical and economic impacts, such as, decreasing prolonged hospitalization and associated costs by shortening overall surgery duration.

DETAILED DESCRIPTION:
This is a non-interventional prospective chart review evaluating the clinical utility of SLND for detecting nodal metastasis of early stage endometrial cancer through data collection.

Patients who are scheduled to undergo standard-of-care (SOC) surgical staging for EC (sentinel lymph node dissection (SLND) via laparotomy, laparoscopy or robotic surgery, ±hysterectomy, ±bilateral salpingo-oophorectomy (BSO)) (pelvic and paraaortic lymphadenectomy may (or may not) also be performed in addition to SLND) will be approached for consent. After these patients have completed the above SOC surgical procedures, research staff will review and collect data from their medical charts. For the subset of these patients who are found, during their SOC surgery, to have positive nodes, research staff will continue to review and collect data from their medical charts after their standard of care follow-up visits with their oncologist

All of the patients enrolled on this trial are those who were scheduled to have their sentinel lymph nodes (SLN) removed; that is, all patients enrolled on this trial were consented by the research team because they were already scheduled to undergo sentinel lymph node dissection (SLND) via laparotomy, laparoscopy or robotic surgery, ±hysterectomy, ±bilateral salpingo-oophorectomy (BSO)). As part of this same SOC surgery, some of these patients also may have undergone pelvic and paraaortic lymphadenectomy in addition to SLND.

Within the research database built for this study, patients will be classified into risk strata (either low or high risk EC) as per the Modified Mayo Criteria. This classification will be partly based on the SOC post-surgical International Federation of Gynecology and Obstetrics (FIGO) staging. To establish progression-free survival (PFS) and overall survival (OS), research staff will intermittently perform medical chart reviews for only those patients with nodal metastasis for a minimum of 2 years (maximum of 6 years).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically and/or cytologically confirmed endometrial cancer.
2. Clinically apparent early stage endometrial cancer (i.e. disease confined to the uterus on preoperative work up).
3. Patient has already scheduled an SLND surgery with treating physician.
4. Females aged 18 years or older.
5. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with lymphadenopathy and/or evidence of metastases, either clinically palpable and/or on preoperative radiological imaging.
2. Any preoperative adjuvant therapy for endometrial cancer (e.g. prior pelvic/abdominal radiotherapy (RT), chemotherapy, or retroperitoneal surgery).
3. Patients may not be receiving any investigational agents.
4. Pregnant or breastfeeding patients.
5. Central Nervous System (CNS) restrictions (i.e. brain metastases).
6. Any uncontrolled, intercurrent illness including but not limited to concomitant cancer, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
7. Any serious medical or psychiatric illness/condition.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Due to the nature of the disease under investigation, only women are eligible to participate in this trial. Women of all races and ethnicities may participate in this research study.
Study Population: All of the patients enrolled on this trial are those who were scheduled to have their sentinel lymph nodes (SLN) removed standard of care.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2016-07-28 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
SLND Positivity Rate in Study Participants | Up to 6 years
  The rate of SLND positivity rate overall and by risk group in patients with clinically apparent early-stage EC. EC patients will be classified as high or low risk group based on the modified Mayo Criteria (Mariani A 2008, Milam 2012).

SECONDARY OUTCOMES:
Rate of NPV and FNPV of the SLND Procedure in Study Participants Who Undergo Partial or Full Lymphadenectomy. | Up to 6 years
  The rate of the negative predictive value (NPV) and its complement the false negative predictive value (FNPV) rate of the SLND procedure in the subset of patients who also undergo partial or full lymphadenectomy. Negative Predictive Value (NPV) will be calculated by dividing the number of true negatives by the total number of patients with a negative SLN (false negatives and true negatives. False Negative Predictive Value (FNPV) rate will be calculated as the number false negatives divided by all patients without nodal metastasis (the number of false negatives and true negatives). FNPV rate is also known as the False Omission Rate (FOR); FNPV is the complement of NPV.
Proportion of Types of Lymph Node Metastases Described by SLND in Study Participants | Up to 6 years
  Proportion of type(s) of lymph node metastases (isolated tumor cells (ITC), micrometastases, or macrometastases) described by SLND in true positive (TP) and false negative (FN) patients. True positives (TPs) are those patients with positive SLN who also have nodal metastasis. False negatives (FNs) are those patients with negative SLN who have nodal metastasis.
Comparison of Nodal Positivity Rates and the Pathologic Protocol for Sentinel Lymph Node Biopsies. | Up to 6 years
  The investigators will compare nodal positivity rates using sentinel lymph node biopsies, and the pathologic protocol for sentinel lymph node biopsies. Positivity rates will be correlated to traditional pathologic factors, including grade, depth of invasion, lymphovascular space invasion, cervical involvement, and histology. Once this information is collected, the investigators will try to assess rates of sentinel lymph node positivity, and its association with these factors.
Rate of Progression-Free Survival in Study Participants With Nodal Metastasis | Up to 6 years
  The rate of progression-free survival (PFS) in patients with nodal metastasis. Progression-Free Survival is defined as the length of time from the date of first dose of study treatment until date of disease progression or death due to any cause, whichever comes first.
Rate of Overall Survival in Study Participants With Nodal Metastasis | Up to 6 years
  The rate of overall survival (OS) in patients with nodal metastasis. Overall survival is defined as the length of time from either the date of first dose of study treatment until death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Slomovitz, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No